CLINICAL TRIAL: NCT02479646
Title: Single Center, Randomized, Double-blind, 3-Period, 3-Treatments, 3-Way Crossover Pharmacokinetics (PK)/Pharmacodynamics (PD) Trial to Assess PK, PD,Safety and Tolerability of MYL-1401H After Single Subcutaneous Injection at One Dose Level (2 mg) Comparing to an EU and US Marketed Drug Product (Neulasta®) in Healthy Volunteers.
Brief Title: Pharmacokinetic / Pharmacodynamic Study Comparing MYL-1401H, EU-sourced Neulasta and US-licensed Neulasta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MYL-1401H-1001; 2014-002229-37 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-24 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: Pegfilgrastim; G-CSF; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — MYL-1401H; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): MYL-1401H: single subcutaneous injection (2mg)
  Interventions: Biological: MYL-1401H
- Treatment B (Active Comparator): EU-Neulasta: single subcutaneous injection (2mg)
  Interventions: Biological: EU-Neulasta
- Treatment C (Active Comparator): US-Neulasta: single subcutaneous injection (2mg)
  Interventions: Biological: US-Neulasta

INTERVENTIONS:
Biological: MYL-1401H
  Other Names: Recombinant human granulocyte colony-stimulating factor (G-CSF); Pegfilgrastim
  Arms: Treatment A
Biological: EU-Neulasta
  Other Names: Recombinant human granulocyte colony-stimulating factor (G-CSF); Pegfilgrastim
  Arms: Treatment B
Biological: US-Neulasta
  Other Names: Recombinant human granulocyte colony-stimulating factor (G-CSF); Pegfilgrastim
  Arms: Treatment C

SUMMARY:
This is a single center, double-blind, randomized, comparative pharmacokinetic and pharmacodynamic study of MYL-1401H and Neulasta (from EU and US source) in Normal Healthy Volunteers.

DETAILED DESCRIPTION:
After successful screening, each subjects will be randomly allocated to one of the following six possible sequences, according a 1:1:1:1:1:1 randomization scheme:

Sequence_1: Treatment A -> Treatment B -> Treatment C ; Sequence_2: Treatment A -> Treatment C -> Treatment B ; Sequence_3: Treatment B -> Treatment A -> Treatment C ; Sequence_4: Treatment B -> Treatment C -> Treatment A ; Sequence_5: Treatment C -> Treatment A -> Treatment B ; Sequence_6: Treatment C -> Treatment B -> Treatment A ;

In study Period 1, Subjects will be administered MYL-1401H (Treatment A), EU-Neulasta(Treatment B) or US-Neulasta (Treatment C).

After the 1st crossover, subjects will enter Study period 2 and will receive one of the remaining alternate treatments.

After the 2nd crossover, subjects will enter Study period 3 and will receive the other alternate treatment.

The washout between drug administrations is at least 4 weeks. Final follow-up visit is scheduled 4 weeks after the last study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Weight: ≥60 kg.
* Body mass index (BMI): 19.0-30.0 kg/m2
* Vital signs showing no clinically relevant deviations.
* Computerized 12-lead ECG recording without signs of clinically relevant pathology.
* Non-smoker or light smoker
* Ability and willingness to abstain from alcohol from 48 hours prior to each admission to the clinical research center and prior to ambulatory visits, and during the stays in the clinic.
* Fertile males and females participating in heterosexual sexual relations: willingness to use adequate contraception from screening until 90 days after the follow up visit
* Females must not be lactating and must have a negative pregnancy test at screening and each admission.
* ANC, total leukocyte count, platelet count, hematocrit and hemoglobin results within the reference ranges.
* All other values for hematology and for clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Principal Investigator

Other protocol specific inclusion/exclusion criteria may apply

Exclusion Criteria:

* Unable to follow protocol instructions in the opinion of the Principal Investigator.
* Any past or concurrent medical conditions that potentially increase the subject's risks or affect the evaluation of any study results. Examples of these include medical history with evidence of clinically relevant pathology (e.g. sickle cell disorders, spleen pathologies, hematologic malignancies or myelodysplastic disorders, and pulmonary illnesses such as ARDS, interstitial pneumonia, pulmonary edema, pulmonary infiltrates and pulmonary fibrosis) and history of relevant drug and/or food allergies.
* Known history of previous exposure to filgrastim, pegfilgrastim, granulocyte colony stimulating factor (GCSF) or any analogue of these.
* Hypersensitivity to the constituents of Neulasta® (sorbitol E420, polysorbate 20 and acetate or acetic acid) or hypersensitivity to E. coli derived proteins.
* Any infection, cough or fever within 1 week prior to first study drug administration.
* Fructose intolerance.
* First degree relatives with hematological malignancy.
* Treatment with non-topical medications within 5 days prior to first admission to the clinical research center, with the exception of hormonal contraceptives, multivitamins, vitamin C, food supplements and a limited amount of paracetamol (acetaminophen), which may be used throughout the study.
* Participation in a drug study within 60 days prior to study drug administration.
* Donation or loss of more than 500 mL of blood over a period of 60 days prior to study drug administration. Donation of more than 1.5 L of blood (for men) / more than 1.0 L of blood (for women) in the 10 months preceding the start of this study.
* History of alcohol abuse or drug addiction
* Regular intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits).
* Positive drug screen (opiates, methadone, cocaine, amphetamines (including ecstasy), cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol).
* Positive screen on hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or anti-human immunodeficiency virus (HIV) 1/2 antibodies.

Other protocol specific inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Area under the curve above baseline of ANC [ANC_AUC(0-tlast)] | Day 1 (0.5, 1, 2, 4, 6, 8, 10, 12, 20 h), and on Days 2, 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29
Pharmacodynamics: Maximum change from baseline in absolute neutrophil count (ANC); ANC_Cmax | Day 1 (0.5, 1, 2, 4, 6, 8, 10, 12, 20 h), Days 2, 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29
Area under the serum concentration-time curve (AUC0-inf) of Pegfilgrastim | Day 1 (0.5, 1, 2, 4, 6, 8, 10, 12, 20 h), Days 2, 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29
  Pharmacokinetics as measured by total AUC after extrapolation from time t to time infinity
Maximum Serum Concentration (Cmax) of pegfilgrastim | Day 1 (0.5, 1, 2, 4, 6, 8, 10, 12, 20 h), Days 2, 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29
  Pharmacokinetics as measured by peak serum concentration of Pegfilgrastim

SECONDARY OUTCOMES:
Frequency of Adverse Events | Daily until Day 9, then on Day 12, 15, 22 of each study period, and at follow-up visit (day 84).
  Safety as measured by incidence of Adverse Events
Safety Variable - Tolerability as measured by Injection Site reactions | Daily until Day 5 of each period
  Tolerability as measured by Injection Site reactions
Safety Variable - Immunogenicity as measured by presence of Anti Drug Antibodies | Day 1 each period and at follow-up (Day 84)
  Immunogenicity as measured by presence of Anti Drug Antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Renger Tiessen, MD, PhD, Principal Investigator — PRA Health Sciences; Fausto Berti, Study Director — Mylan GmbH
Locations (1):
- PRA Health Sciences - Early Development Services, Zuidlaren, Netherlands